CLINICAL TRIAL: NCT03559920
Title: The Optimal Dose of Sevoflurane Via Anaconda® in Post-operative Patient Underwent Head & Neck Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0065
Record Dates: First submitted 2018-06-01; First posted 2018-06-18 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Patients Who Needs Sedation After Head & Neck Surgery
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Experimental): Patients who are sedated using sevoflurane
  Interventions: Drug: Sedate using sevoflurane via anesthetic conserving device(ACD, Anaconda®) after surgery
- Intravenous sedation group (Active Comparator): Patients who are sedated using propofol
  Interventions: Drug: Sedate using propofol.

INTERVENTIONS:
Drug: Sedate using sevoflurane via anesthetic conserving device(ACD, Anaconda®) after surgery — The investigators sedate the patients in the ICU for several days after head & neck surgery using sevoflurane via anesthetic conserving device in sevoflurane group.
  Arms: Sevoflurane group
Drug: Sedate using propofol. — Retrospectively, the investigators compare the sevoflurane group with intravenous sedation group using propofol.
  Arms: Intravenous sedation group

SUMMARY:
Sedation in the ICUs is very common. There is no ideal sedative yet, so research has been conducted to replace propofol and midazolam, which are the most commonly used sedatives in ICUs, by inhalation anesthetics. The investigators will sedate the patients who undergo head & neck surgery with tracheostomy for several days using sevoflurane, a kind of inhalation agent, via anesthetic conserving device.

The objective of this study is to confirm the end-tidal sevoflurane concentration for inducing moderate sedation (RASS -2~-3). In addition, the investigators compare the volatile sedation with the IV(intravenous) sedation to see if the volatile sedation could reduce the amount of post-operative opioid consumption.

* RASS: Richmond Agitation-Sedation Scale
* RASS: Richmond Agitation-Sedation Scale

DETAILED DESCRIPTION:
When patients, who need mechanical ventilation for several days after head & neck surgery, enters the ICU, the investigators induce moderate sedation (RASS -2~-3). End-tidal sevoflurane (etSEVO) concentration is adjusted to 0.5Vol% within 30 minutes. Sedation level is evaluated every 5 minutes. After 30 minutes, the investigators check that the sedation goal is achieved.

Following the up & down method, if the moderate sedation (RASS -2~-3) or the deep sedation (RASS -4~-5) is achieved at the etSEVO concentration of 0.5vol% after 30 minutes of sedation, the next patient's target etSEVO concentration is reduced to 0.4vol%. On the contrary to this, if only light sedation (RASS above -1) is achieved, the next patient's target etSEVO is increased to 0.6vol%. This process is repeated to find the appropriate etSEVO concentration at the beginning of sedation, which induces sedation of RASS -2~-3.

In retrospective analysis, the investigators compared the prospective study group with propofol intravenous sedation group.

* RASS: Richmond Agitation-Sedation Scale

ELIGIBILITY:
Inclusion Criteria:

* Patients who needs sedation in the ICU for several days after head & neck surgery
* ASA class I~III
* Adult patients over 20 years old
* Patients who can read and understand the informed consent

Exclusion Criteria:

* Patients who do not agree to participate in the study
* Past history or Family history of malignant hyperthermia
* End stage renal disease (eGFR<30 or dialysis)
* Moderate to severe liver disease (AST, ALT > 200IU/L)
* Pregnant women
* Patients who cannot read and understand the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Optimal end-tidal sevoflurane concentration to induce moderate sedation of RASS -2~-3 in patients who undergo head & neck surgery with tracheostomy | After the first 30 minutes after sedation with sevoflurane via anesthetic conserving device
  Investigators will find the initial concentration of sevoflurane for proper sedation by the Dixon's up and down method.

SECONDARY OUTCOMES:
Compare the sevoflurane group and the intravenous sedation group: Compare the ICU stay | within the 3 days (plus of minus 3 days) after surgery
Compare the sevoflurane group and the intravenous sedation group: Compare the hospital day | within the 3 days (plus of minus 3 days) after surgery
Compare the sevoflurane group and the intravenous sedation group: Compare the incidence of delirium, hypotension | within the 3 days (plus of minus 3 days) after surgery
Compare the sevoflurane group and the intravenous sedation group: Compare the remifentanil infusion dose | within the 3 days (plus of minus 3 days) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea